CLINICAL TRIAL: NCT04123366
Title: A Phase 2 Study of Olaparib in Combination With Pembrolizumab in Participants With Previously Treated, Homologous Recombination Repair Mutation (HRRm) and/or Homologous Recombination Deficiency (HRD)-Positive Advanced Cancer
Brief Title: Study of Olaparib (MK-7339) in Combination With Pembrolizumab (MK-3475) in the Treatment of Homologous Recombination Repair Mutation (HRRm) and/or Homologous Recombination Deficiency (HRD)-Positive Advanced Cancer (MK-7339-007/KEYLYNK-007)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7339-007; MK-7339-007 (Other: MSD); KEYLYNK-007 (Other: MSD); jRCT2011200025 (Registry Identifier: jRCT); 2023-503831-17 (Registry Identifier: EU CT); U1111-1288-1642 (Registry Identifier: UTN); 2019-001745-40 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — olaparib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib+Pembrolizumab (Experimental): Participants receive olaparib 300 mg via oral tablet 2 times each day PLUS pembrolizumab 200 mg via intravenous infusion on Day 1 of each 21-day cycle. Participants may receive olaparib+pembrolizumab for up to approximately 2 years.
  Interventions: Drug: Olaparib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Olaparib — Oral tablet
  Other Names: MK-7339; LYNPARZA®
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of treatment with olaparib (MK-7339) in combination with pembrolizumab (MK-3475) in adults with previously treated, advanced (metastatic and/or unresectable) Homologous Recombination Repair Mutation (HRRm) and/or Homologous Recombination Deficiency (HRD)-positive solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced (metastatic and/or unresectable) solid tumor (except breast or ovarian cancers whose tumor has a germline or somatic BRCA mutation) that is not eligible for curative treatment and for which standard of care therapy has failed. Participants must have progressed on or be intolerant to standard of care therapies that are known to provide clinical benefit. There is no limit on the number of prior treatment regimens.
* Has either centrally-confirmed known or suspected deleterious mutations in ≥1 of the specified 15 genes involved in HRR or centrally-confirmed HRD based on the Lynparza HRR-HRD assay.
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology and confirmed in real time by blinded independent central review (BICR). BICR must confirm the presence of radiologically measurable disease per RECIST 1.1 for the participant to be eligible for the study.
* Has a life expectancy of ≥3 months.
* Must have had CR or PR while on the last treatment with prior cisplatin or carboplatin, or if received only oxaliplatin had CR, PR, or stable disease (SD) while on the last treatment with prior oxaliplatin (either as monotherapy or in combination) for advanced (metastatic and/or unresectable) solid tumor. Participant must also not have been refractory to prior platinum-containing therapy.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1, as assessed within 3 days of study treatment initiation.
* Male participants must agree to use contraception during the treatment period and for ≥90 days (3 months) after the last dose of olaparib and refrain from donating sperm during this period.
* Female participants must not be pregnant or breastfeeding, and ≥1 of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP who agrees to use contraception during the treatment period and for ≥120 days (3 months) after the last dose of pembrolizumab and 180 days (6 months) after the last dose of olaparib, has a highly sensitive pregnancy test within 24 hours for urine or within 72 hours for serum before the first dose of study intervention, and abstains from breastfeeding during the study intervention period and for at least 120 days after the last dose of the study intervention.
* Has adequate organ function

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal carcinoma in situ, or cervical carcinoma in situ that has undergone potentially curative therapy are not excluded.
* Has a history of non-infectious pneumonitis/interstitial lung disease that required treatment with steroids or currently has pneumonitis/interstitial lung disease.
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active infection requiring systemic therapy.
* Has active tuberculosis (Bacillus tuberculosis [TB]).
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing >10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has received colony-stimulating factors (e.g. granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study treatment.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active hepatitis B or hepatitis C.
* Is unable to swallow orally administered medication or has a gastrointestinal (GI) disorder affecting absorption (e.g. gastrectomy, partial bowel obstruction, malabsorption).
* Has received prior therapy with an anti-programmed death-1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), or anti-programmed death-ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40 [Tumor necrosis factor receptor superfamily, member 4 (TNFRSF4)], CD137 [tumor necrosis factor receptor superfamily member 9 (TNFRSF9)]).
* Has received prior therapy with olaparib or with any other polyadenosine 5' diphosphoribose (poly[ADP ribose]) polymerization (PARP) inhibitor.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to administration of study treatment.
* Must have recovered from all adverse events (AEs) due to previous therapies, excluding alopecia, to ≤Grade 1 or Baseline.
* Has a known hypersensitivity to the study treatments and/or any of their excipients.
* Is currently receiving either strong inhibitors of cytochrome P450 (CYP)3A4 (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate inhibitors of CYP3A4 (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 2 weeks.
* Is currently receiving either strong inducers of CYP3A4 (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate inducers of CYP3A4 (e.g. bosentan, efavirenz, modafinil) that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
* Has received previous allogenic bone-marrow transplant or double umbilical cord transplantation (dUCBT).
* Has received a whole blood transfusion in the last 120 days prior to entry to the study.
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Is currently enrolled in and receiving study therapy, was enrolled in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks (28 days) of the first dose of study treatment.
* The presence of uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fredericia [QTcF] prolongation >500 msec, electrolyte disturbances), or participant has congenital long QT syndrome.
* Has either had major surgery within 2 weeks of starting study treatment or has not recovered from any effects of any major surgery.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Has had an allogenic tissue/solid tumor organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-07-23 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or Prostate Cancer Working Group (PCWG)-modified RECIST 1.1 in Biomarker Subgroups | Up to ~3 years
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The ORR for all participants will be presented by biomarker subgroup.

SECONDARY OUTCOMES:
Duration of Response (DOR) as Assessed by RECIST 1.1 or PCWG-modified RECIST 1.1 in Biomarker Subgroups | Up to ~3 years
  For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR for all participants who experience a CR or PR will be presented by biomarker subgroup.
Progression-Free Survival (PFS) as Assessed by RECIST 1.1 or PCWG-modified RECIST 1.1 in Biomarker Subgroups | Up to ~3 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more lesions is also considered PD. The PFS for all participants will be presented by biomarker subgroup.
Overall Survival (OS) in Biomarker Subgroups | Up to ~3 years
  OS is the time from randomization to death due to any cause. The OS for all participants will be presented by biomarker subgroup.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~3 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to ~3 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment will be presented.
Objective Response Rate (ORR) Based on Tumor Biomarker Status as Assessed by RECIST 1.1 or PCWG-modified RECIST 1.1 in Additional Biomarker Subpopulations | Up to ~3 years
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR will be presented by biomarker subpopulation.
Duration of Response (DOR) Based on Tumor Biomarker Status as Assessed by RECIST 1.1 or PCWG-modified RECIST 1.1 in Additional Biomarker Subpopulations | Up to ~3 years
  For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR for all participants who experience a CR or PR will be presented by biomarker subpopulation.
Progression-Free Survival (PFS) Based on Tumor Biomarker Status as Assessed by RECIST 1.1 or PCWG-modified RECIST 1.1 in Additional Biomarker Subpopulations | Up to ~3 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more lesions is also considered PD. PFS will be presented by biomarker subpopulation.
Overall Survival (OS) in Additional Biomarker Subpopulations | Up to ~3 years
  OS is the time from randomization to death due to any cause. OS will be presented by biomarker subpopulation.
Number of Participants with Cancer Antigen-125 (CA-125) Level of ≥2 × Upper Limit of Normal (ULN) Among Participants with Ovarian Cancer | Up to ~3 years
  The number of participants who have ovarian cancer and have a CA-125 level ≥2 × upper limit of normal (ULN) at 2 different assessments that are measured at least 1 week apart will be presented.
Number of Participants with Cancer Antigen-125 (CA-125) Level ≥2 × Nadir (Lowest) Value Among Participants with Ovarian Cancer Who Had Elevated CA-125 Levels ≥ULN at Baseline | Up to ~3 years
  The number of participants who have ovarian cancer with an elevated CA-125 level ≥ ULN at Baseline and have a CA-125 level ≥2 × the nadir (lowest) value at 2 different assessments that are measured at least 1 week apart will be presented.
Number of Participants with a Change from Baseline in Prostate-Specific Antigen (PSA) Level of ≥50% Among Participants with Prostate Cancer | Up to ~3 years
  A PSA response is defined as a reduction in the PSA level of ≥50% from Baseline measured at 2 different times at least 3 weeks apart. The number of participants who have prostate cancer and have a change from Baseline in PSA level ≥50% will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (135):
- United States (21):
  - The Kirklin Clinic ( Site 0086), Birmingham, Alabama
  - Banner MD Anderson Cancer Center ( Site 0049), Gilbert, Arizona
  - UC Davis Comprehensive Cancer Center ( Site 0039), Sacramento, California
  - San Francisco Oncology Associates ( Site 0085), San Francisco, California
  - University of California San Francisco ( Site 0015), San Francisco, California
  - Banner MD Anderson Cancer Center ( Site 0092), Greeley, Colorado
  - University of Florida ( Site 0078), Gainesville, Florida
  - Winship Cancer Institute of Emory University ( Site 0057), Atlanta, Georgia
  - Northeast Georgia Medical Center ( Site 0026), Gainesville, Georgia
  - Northwest Georgia Oncology Centers PC ( Site 0047), Marietta, Georgia
  - Norton Cancer Institute - St. Matthews ( Site 0024), Louisville, Kentucky
  - Atlantic Health System ( Site 0046), Summit, New Jersey
  - New York Cancer and Blood Specialists-Research Department ( Site 0080), Port Jefferson Station, New York
  - University Hospitals Cleveland Medical Center ( Site 0016), Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center ( Site 0050), Oklahoma City, Oklahoma
  - Parkland Health & Hospital System ( Site 0091), Dallas, Texas
  - University of Texas, Southwestern Medical Center ( Site 0004), Dallas, Texas
  - University of Texas-MD Anderson Cancer Center ( Site 0087), Houston, Texas
  - Utah Cancer Specialists ( Site 0038), West Valley City, Utah
  - Inova Schar Cancer Institute ( Site 0008), Fairfax, Virginia
  - Northwest Medical Specialties, PLLC ( Site 0007), Tacoma, Washington
- Argentina (5):
  - Fundacion CIDEA ( Site 2704), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 2705), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra De Salvo ( Site 2702), Buenos Aires
  - CEMIC ( Site 2701), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 2703), La Rioja
- Australia (4):
  - Blacktown Hospital ( Site 2202), Blacktown, New South Wales
  - Tasman Oncology Research Pty Ltd ( Site 2203), Southport, Queensland
  - Monash Medical Centre ( Site 2205), Clayton, Victoria
  - Linear Clinical Research Ltd ( Site 2206), Nedlands, Western Australia
- Canada (3):
  - BC Cancer-Vancouver Center ( Site 0203), Vancouver, British Columbia
  - Moncton Hospital - Horizon Health Network ( Site 0206), Moncton, New Brunswick
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0201), Montreal, Quebec
- Colombia (5):
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 2902), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 2900), Barranquilla, Atlántico
  - Fundacion Cardiovascular de Colombia ( Site 2907), Piedecuesta, Santander Department
  - Hemato Oncologos S.A. ( Site 2910), Cali, Valle del Cauca Department
  - Fundacion Valle del Lili ( Site 2909), Cali, Valle del Cauca Department
- France (5):
  - CHU Jean Minjoz ( Site 0606), Besançon, Doubs
  - Institut du Cancer de Montpellier ( Site 0610), Montpellier, Herault
  - Centre Henri Becquerel ( Site 0607), Rouen, Seine-Maritime
  - Institut Gustave Roussy ( Site 0602), Villejuif, Val-de-Marne
  - CHD Vendee ( Site 0604), La Roche-sur-Yon, Vendee
- Germany (3):
  - Universitaetsklinik der Ludwig-Maximilians-Universitaet Muenchen ( Site 0906), Munich, Bavaria
  - Universitaetsklinik Koeln ( Site 0903), Cologne, North Rhine-Westphalia
  - Charite-Universitaetsmedizin Berlin-Campus Benjamin Franklin ( Site 0902), Berlin
- Guatemala (5):
  - Oncologika S.A. ( Site 3003), Guatemala City
  - Grupo Angeles SA ( Site 3004), Guatemala City
  - Sanatorio Nuestra Senora del Pilar ( Site 3006), Guatemala City
  - Medi-K Cayala ( Site 3005), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 3002), Quetzaltenango
- Israel (6):
  - Rambam Health Care Campus-Oncology Division ( Site 0801), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0802), Jerusalem
  - Meir Medical Center ( Site 0804), Kfar Saba
  - Rabin Medical Center ( Site 0806), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0800), Ramat Gan
  - Sourasky Medical Center ( Site 0805), Tel Aviv
- Italy (4):
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 0703), Modena, Emilia-Romagna
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0700), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0705), Napoli
  - Azienda Ospedaliera Universitaria Senese ( Site 0704), Siena
- Japan (7):
  - Aichi Cancer Center Hospital ( Site 2504), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2500), Kashiwa, Chiba
  - Hokkaido University Hospital ( Site 2502), Sapporo, Hokkaido
  - Kyushu University Hospital ( Site 2506), Fukuoka
  - Okayama University Hospital ( Site 2505), Okayama
  - National Cancer Center Hospital ( Site 2501), Tokyo
  - Japanese Foundation for Cancer Research ( Site 2503), Tokyo
- Latvia (4):
  - Daugavpils Regional Hospital ( Site 2104), Daugavpils
  - Liepaja Regional Hospital ( Site 2101), Liepāja
  - Riga East Clinical University Hospital ( Site 2103), Riga
  - P. Stradina Clinical University Hospital ( Site 2102), Riga
- Mexico (7):
  - Preparaciones Oncologicas ( Site 3102), León, Guanajuato
  - Unidad Biomedica Avanzada Monterrey S. A. ( Site 3108), Monterrey, Nuevo León
  - Centro Medico Zambrano Hellion ( Site 3105), San Pedro Garza García, Nuevo León
  - Hospital H+ Queretaro ( Site 3104), Querétaro City, Querétaro
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 3101), Madero, Tamaulipas
  - CRYPTEX Investigacion Clinica S.A. de C.V. ( Site 3103), Mexico City
  - Clinica Integral Internacional de Oncologia S. de R.L. de C.V. ( Site 3107), Puebla City
- Peru (8):
  - Hospital Nacional Carlos Alberto Seguin Escobedo ESSALUD ( Site 3206), Arequipa, Ariqipa
  - Hospital Nacional Daniel Alcides Carrion ( Site 3207), Bellavista, Qallaw
  - Hospital Nacional Adolfo Guevara Velasco ( Site 3205), Cuzco, Qusqu
  - Oncosalud ( Site 3200), Lima
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 3201), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 3208), Lima
  - Clinica San Gabriel ( Site 3202), Lima
  - Hospital Nacional Cayetano Heredia ( Site 3203), Lima
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 1809), Gdansk, Pomeranian Voivodeship
- Puerto Rico (4):
  - Hematology and Oncology Institute ( Site 0504), Manatí
  - Ad-Vance Medical Research LLC ( Site 0505), Ponce
  - Pan American Center for Oncology Trials LLC ( Site 0501), Rio Piedras
  - FDI Clinical Research ( Site 0500), San Juan
- Romania (5):
  - Spitalul Judetean de Urgenta Alba Iulia ( Site 1107), Alba Iulia, Alba
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1101), Cluj-Napoca, Cluj
  - Medisprof ( Site 1102), Cluj-Napoca, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1103), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 1104), Timișoara, Timiș County
- South Africa (6):
  - Universitas Annex National Hospital ( Site 1902), Bloemfontein, Free State
  - Wits Clinical Research ( Site 1906), Parktown-Johannesburg, Gauteng
  - Mary Potter Oncology Centre, Little Company of Mary Hospital ( Site 1900), Pretoria, Gauteng
  - Vaal Triangle Oncology Centre ( Site 1905), Vereeniging, Gauteng
  - The Oncology Centre ( Site 1904), Durban, KwaZulu-Natal
  - Cancercare Rondebosch Oncology ( Site 1901), Rondebosch, Western Cape
- South Korea (4):
  - Seoul National University Bundang Hospital ( Site 2403), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 2402), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2400), Seoul
  - Samsung Medical Center ( Site 2401), Seoul
- Spain (3):
  - Hospital Quiron de Madrid ( Site 1301), Pozuelo de Alarcón, Madrid
  - Hospital Clinic i Provincial ( Site 1302), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1300), Madrid
- Sweden (3):
  - Skanes Universitetssjukhus Lund. ( Site 2001), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 2000), Solna, Stockholm County
  - Akademiska Sjukhuset ( Site 2002), Uppsala, Uppsala County
- Turkey (Türkiye) (11):
  - Baskent University Adana Training Hospital ( Site 1509), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1502), Ankara
  - Gazi Universitesi Tip Fakultesi ( Site 1507), Ankara
  - Ankara Sehir Hastanesi ( Site 1508), Ankara
  - Akdeniz Universitesi Tıp Fakultesi ( Site 1503), Antalya
  - Trakya University Medical Faculty Balkan Oncology Hospital ( Site 1500), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1504), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi ( Site 1505), Istanbul
  - Ege Universitesi Tip Fakultesi Tulay Aktas Onkoloji Hastanesi ( Site 1501), Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi ( Site 1510), Konya
  - Inonu Universitesi Medical Fakultesi ( Site 1506), Malatya
- Ukraine (10):
  - Cherkasy Regional Oncology Dispensary ( Site 1702), Cherkasy, Cherkasy Oblast
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council ( Site 1700), Dnipro, Dnipropetrovsk Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical On-Department for daily treated patient (, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1704), Kharkiv, Kharkivs’ka Oblast’
  - Khmelnitskiy Regional Onkology Dispensary ( Site 1705), Khmelnitskiy, Khmelnytskyi Oblast
  - Kirovograd Regional oncology Dispensary ( Site 1716), Kropyvnytsky, Kirovohrad Oblast
  - Medical Centre Consilium Medical ( Site 1712), Kyiv, Kyivska Oblast
  - Podillya Regional Center of Oncology ( Site 1708), Vinnytsia, Vinnytsia Oblast
  - Medical center of the Limited Liability Company Yulis ( Site 1714), Zaporizhzhia, Zaporizhzhia Oblast
  - Zhytomyr Regional Oncology Center ( Site 1710), Zhytomyr, Zhytomyr Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Cannon TL, Randall JN BA, Sokol ES, Alexander SM, Wadlow RC, Winer AA, Barnett DM, Rayes DL BS, Nimeiri HS, McGregor KA. Concurrent BRAFV600E and BRCA Mutations in MSS Metastatic Colorectal Cancer: Prevalence and Case Series of mCRC patients with prolonged OS. Cancer Treat Res Commun. 2022;32:100569. doi: 10.1016/j.ctarc.2022.100569. Epub 2022 Apr 30. PMID 35567913
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26263&tenant=MT_MSD_9011